CLINICAL TRIAL: NCT04840225
Title: Anæmi Hos Patienter Med infektiøs Endokarditis - Karakteristik og Mekanismer (ANIE)
Brief Title: Anemia in Patients With Endocarditis
Acronym: ANIE
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mia Pries-Heje, MD, Rigshospitalet, Denmark
Other Study IDs: H-20044379
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Anemia; Endocarditis, Bacterial
MeSH Terms: conditions — Anemia; Endocarditis, Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Endocarditis: 100 patients diagnosed with infectious endocarditis according to DUKE criteria. Detailed characterization of inflammation, anemia and markers of iron hemostatis will be made at diagnosis and followed undtill 6 months after discharge.
  Interventions: Other: Measurement of biomarkers for inflammation and anemia
- TAVI/TEVAR patietns: 30 patients undergoing elektive TAVI/TEVAR procedures. Detailed characterization of inflammation, anemia and markers of iron hemostatis will be made at directly prior to procedure and followed undtill 3 months after discharge.
  Interventions: Other: Measurement of biomarkers for inflammation and anemia
- Patients with bacterial infections without endocarditis: 30 patients diagnosed with with bacterial infections, without endocarditis. Detailed characterization of inflammation, anemia and markers of iron hemostatis will be made at diagnosis and followed undtill 3 months after discharge.
  Interventions: Other: Measurement of biomarkers for inflammation and anemia
- Healthy blood donors: Detailed characterization of inflammation, anemia and markers of iron hemostatis will be made at directly prior to blood donation and approximately 1 week after blood donations
  Interventions: Other: Measurement of biomarkers for inflammation and anemia

INTERVENTIONS:
Other: Measurement of biomarkers for inflammation and anemia — Measurement of biomarkers for inflammation and anemia, in addition to standart clinical measurements

SUMMARY:
Prospective study of prevalence and deep charecterization of anemia in patients with endocarditis from diagnosis undtill 6 months after discharge.

DETAILED DESCRIPTION:
Anemia is an adverse prognostic marker in both cardiac diseases and infectious diseases. In patients with bacterial endocarditis (IE), anemia has a prevalence of 55-80%. In a sub-study to our POET I trial (RCT with 400 patients with IE, published in NEJM 2019), preliminary data show a 5-fold increased risk of death within 6 months and 2-fold increased risk after 3 years, in non-surgically treated patients with hemoglobin <6.2mmol/L, compared to patients with no or mild anemia. Intensified treatment of anemia through e.g. intravenous iron infusions, in combination with erythrocyte stimulating agents or new treatments for anemia of inflammation, such as IL-6 inhibitors, could possibly improve outcome for patients with IE.

This study - ANIE - is a prospective study, aiming at further deep-characterizing of anemia in patients with IE, and associated outcomes. Degree of anemia of inflammation (AI) and iron-deficiency anemia during hospitalization and time to recovery will be assessed. Blood samples from 100 patients with IE will be collected during hospitalization and 3 months after discharge, i.e. also during expected recovery. Samples will be analyzed for standard markers of anemia and inflammation, as well as novel biomarkers for AI, such as IL-6, soluble transferrin receptor, erythroferrone and hepcidin. The sample size calculation is based on the assumption that the prevalence of AI is 50%, with a confidence interval of 95% and a margin of error of <10%. Comparisons will be made to patients with other infections and patients with pure inflammation (TAVI and TEVAR patients) and healthy blood donors.

ANIE is expected to give us an unprecedented insight into disease processes, stages and possible therapeutic targets for anemia in patients with IE.

The results will serve for designing the clinical trial of novel interventions to treat anemia in patients with IE, as a novel means to improve the outcome and reduce the high mortality in these patients.

Anemia is an adverse prognostic marker in both cardiac diseases and infectious diseases. In patients with bacterial endocarditis (IE), anemia has a prevalence of 55-80%. In a sub-study to our POET I trial (RCT with 400 patients with IE, published in NEJM 2019), preliminary data show a 5-fold increased risk of death within 6 months and 2-fold increased risk after 3 years, in non-surgically treated patients with hemoglobin <6.2mmol/L, compared to patients with no or mild anemia. Intensified treatment of anemia through e.g. intravenous iron infusions, in combination with erythrocyte stimulating agents or new treatments for anemia of inflammation, such as IL-6 inhibitors, could possibly improve outcome for patients with IE.

This study - ANIE - is a prospective study, aiming at further deep-characterizing of anemia in patients with IE, and associated outcomes. Degree of anemia of inflammation (AI) and iron-deficiency anemia during hospitalization and time to recovery will be assessed. Blood samples from 100 patients with IE will be collected during hospitalization and 3 months after discharge, i.e. also during expected recovery. Samples will be analyzed for standard markers of anemia and inflammation, as well as novel biomarkers for AI, such as IL-6, soluble transferrin receptor, erythroferrone and hepcidin. The sample size calculation is based on the assumption that the prevalence of AI is 50%, with a confidence interval of 95% and a margin of error of <10%. Comparisons will be made to patients with other infections and patients with pure inflammation (TAVI and TEVAR patients) and healthy blood donors.

ANIE is expected to give us an unprecedented insight into disease processes, stages and possible therapeutic targets for anemia in patients with IE.

The results will serve for designing the clinical trial of novel interventions to treat anemia in patients with IE, as a novel means to improve the outcome and reduce the high mortality in these patients.

ELIGIBILITY:
IE-patients:

Inclusion Criteria:

• Infectious endocarditis, defined by Duke criteria

Exclusion Criteria:

• Known rheumatic disease or immune defect

TAVI/TEVAR patients:

Inclusion Criteria:

• Scheduled for a TAVI/TEVAR procedure

Exclusion criteria:

* Clinical suspicion of infection
* Known rheumatic disease or immune defect

Bacterial patients without IE (short infection):

Inclusion criteria

* Patients admitted with an infection with gram positive bacteria, without IE Exclusion criteria
* Known rheumatic disease or immune defect

Blood donors:

Exclusion criteria:

* Antibiotic treatment within the last 2 months
* Cancer, rheumatic disease or other known inflammatory disease
* Surgery within the last 3 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with IE, 30 undergoing elective TAVI/TECAR, 30 with non-IE bacterial infections and 30 healthy blood donors
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia during hospitalization | From time of diagnosis/intervention untill end of follow-up (up to 6 months from inclusion)
  Diagnosis of anemia through WHO/NCI criteria for anemia and severity of anemia at time of diagnosis, 1-4 weeks after initiation of relevant treatment and up to 6 months after discharge

SECONDARY OUTCOMES:
Prevalence of iron deficiency anemia in patients with IE and relevant controls | From time of diagnosis/intervention untill end of follow-up (up to 6 months from inclusion)
  Determination of the prevalence of iron deficiency anemia through measurements of hemoglobin, markers of anemia and of iron metabolism/stores in blood
Prevalence of anemia due to inflammation in patients with IE and relevant controls | From time of diagnosis/intervention untill end of follow-up (up to 6 months from inclusion)
  Determination of the prevalence of anemia og inflammation through measurements of markers of anemia of inflammation (IL-6 hepcidin, erytroferrone, soluble transferrin receptor)
Time untill resolution of inflammation and anemia in patients with IE and relevant controls | From time of diagnosis/intervention untill end of follow-up (up to 6 months from inclusion)
  Determination of time from start of treatment/intervention until normalization of markers of inflammation and anemia, as well as normalization of erythropoiesis

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Available on reasonable request